CLINICAL TRIAL: NCT06387095
Title: Efficacy of Parasternal Blocks in Cardiovascular Surgery Patients Undergoing Median Sternotomy: Randomized, Controlled Study
Brief Title: Efficacy of Parasternal Blocks in Cardiovascular Surgery Patients Undergoing Median Sternotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, münire deniz, Principal Investigator Medical Doctor, Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/01/756
Record Dates: First submitted 2024-04-04; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Pain
Keywords: postoperative pain; parasternal blocks; chronic pain; acute pain; cabg
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain; Acute Pain

STUDY DESIGN:
Intervention Model Description: randomized controlled
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1. control group (Active Comparator): control group. block will not be applied to this group and the patient's analgesia needs will be provided with patient-controlled analgesia devices.
  Interventions: Procedure: 1. no block
- 2. superficial parasternal plane block group (Active Comparator): superficial parasternal plane block group. superficial paraasternal plane block will be applied to this group. it will be applied to the parasternal region with ultrasound after the patient is intubated. patient-controlled analgesia devices will be used for additional postoperative pain needs.
  Interventions: Procedure: 2. superficial parasternal block
- 3. deep parasternal plane block group (Active Comparator): deep parasternal plane block group. deep paraasternal plane block will be applied to this group. it will be applied to the parasternal region with ultrasound after the patient is intubated. patient-controlled analgesia devices will be used for additional postoperative pain needs.
  Interventions: Procedure: 3. deep parasternal block

INTERVENTIONS:
Procedure: 1. no block — After extubation, patient-controlled analgesia will be applied for 24 hours (with PCA infusion pump device). During the follow-up of the patients in intensive care, extubation times, additional analgesic needs, pain scores; intensive care and hospital discharge times will be recorded.
  Other Names: intravenous analgesia
  Arms: 1. control group
Procedure: 2. superficial parasternal block — After induction, the patient will undergo an ultrasound-guided superficial parasternal plan block. . After extubation, patient-controlled analgesia will be applied for 24 hours (with PCA infusion pump device). During the follow-up of the patients in intensive care, extubation times, additional analgesic needs, pain scores; intensive care and hospital discharge times will be recorded.
  Other Names: intravenous analgesia; regional analjesia
  Arms: 2. superficial parasternal plane block group
Procedure: 3. deep parasternal block — After induction, the patient will undergo an ultrasound-guided deep parasternal plane block. . After extubation, patient-controlled analgesia will be applied for 24 hours (with PCA infusion pump device). During the follow-up of the patients in intensive care, extubation times, additional analgesic needs, pain scores; intensive care and hospital discharge times will be recorded.
  Other Names: intravenous analgesia; regional analjesia
  Arms: 3. deep parasternal plane block group

SUMMARY:
Acute and chronic pain after cardiac surgery is a common problem that negatively affects quality of life. Postoperative pain after cardiac surgery is most intense in the first two days and decreases in the following period. However, postoperative pain with incomplete management in the acute period may become chronic. This may negatively affect the patient's quality of life. Although central blocks such as thoracic epidural and paravertebral blocks are considered the gold standard in analgesia control, the advantages of thoracic plan blocks, which are more superficial due to peroperative heparinisation; coagulation disorders; and procedural difficulties, are undeniable. Thoracic plane blocks, which can also be used in patients receiving anticoagulant and/or antiplatelet therapy, have recently been used for acute pain. The aim of this study was to evaluate the effect of thoracic plane blocks on extubation time, pain scores, intensive care unit (ICU) and hospital stays in patients undergoing median sternotomy.

DETAILED DESCRIPTION:
The study will proceed in three arms. The first group is the control group and will receive total intravenous anaesthesia as infusion after peroperative induction until the patient leaves the operating room. The second group will receive ultrasound-guided parasternal superficial plan block after induction. The third group will receive ultrasound-guided parasternal deep plan block. Extubation times, additional analgesic needs, pain scores, intensive care unit duration and hospital discharge times will be compared in the three groups during intensive care unit follow-up. After extubation, patient-controlled analgesia will be applied for 24 hours (with pca infusion pump device).

ELIGIBILITY:
Inclusion Criteria:

* Performing median sternotomy
* Elective case
* Over 18 years of age; under 80 years of age
* ASA II-III patients

Exclusion Criteria:

* Emergency cases
* Patients undergoing minimally invasive surgery
* Patients with a history of opioid use in the last 30 days
* Redo cases
* Patients with left ventricular ejection fraction less than 30%
* Patients with severe hepatic or renal insufficiency
* Patients with chronic pain before surgery (migraine, fibromyalgia)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
postoperative chronic pain | 6 months
  Determination the effect of parasternal blocks on the incidence for chronic pain at 6 months postoperative period in cardiac surgery. The s-lanss scores of the patients at the 6th postoperative month will be evaluated. The range of the questionnaire is 0-24 and patients with a score above 12 will be considered to have neuropathic pain.

SECONDARY OUTCOMES:
postoperative 24 hours acute pain | 24 hours
  postoperative 24 hours pain of the patients will be evaluated with VAS (visual analogue scale). analgesic needs of the patients in the first 24 hours postoperatively will be calculated as morphine equivalent dose using PCA device. At the end of the 24th hour, BPI (brief pain index) will be evaluated. additional analgesic needs of the patients (NSAID, narcotic), if any, will be recorded. it will be evaluated whether there is a significant difference between the VAS scores, analgesic needs and BPI scores in the first 24 hours pain according to the groups.
extubation time | 24 hours
  Extubation time (defined as the time from admission to intensive care unit until extubation) will be evaluated for differences between the groups.the control group
icu time | 7 days
  The study will look at whether intensive care and hospital discharge times differ between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: munire deniz, Study Director — kosuyolu high education and training center
Locations (1):
- Kosuyolu High Education and Training Hospital, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No